CLINICAL TRIAL: NCT04851457
Title: Safety and Efficacy of Tirofiban in Acute Ischemic Stroke Patients Treated With Mechanical Thrombectomy-A Prospective, Randomized, Controlled, Open-Label, Assessor-Blind, Multicenter Clinical Study
Brief Title: One Pass Tirofiban In Management of Ischemic Stroke Thrombectomy In China
Acronym: OPTIMISTIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Collaborators: Shanghai 6th People's Hospital (Other); Ningbo No. 1 Hospital (Other); Zhangzhou Municipal Hospital of Fujian Province (Other); Shanghai 7th People's Hospital (Other); Jinan Central Hospital (Other); Xuchang Central Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-OPTIMISTIC
Record Dates: First submitted 2021-04-11; First posted 2021-04-20 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Ischemic Stroke
Keywords: Acute Ischemic Stroke; Tirofiban; Mechanical thrombectomy; Revascularisation; Haemorrhage
MeSH Terms: conditions — Ischemic Stroke; Hemorrhage | interventions — Tirofiban

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled, open-Label, assessor-blind, multicenter clinical study
Who Masked: Outcomes Assessor
Masking Description: Images from each study site will be uploaded to the central server and all analyses will be performed by a trained physician at the study coordinating center who is unaware of group assignments. Similarly, follow-up assessments at 90 days after stroke will be conducted by a trained accessor in a blinded manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The participants in the experimental group will receive intravenous tirofiban combined with a standard MT protocol recommended by the current guidelines for the management of AIS
  Interventions: Drug: Intravenous tirofiban combination therapy
- Control group (No Intervention): Patients are treated with MT therapy with no antiplatelet drugs (intravenous or intra-arterial) are administered. Besides, they will receive a standard pharmacological treatment as per current clinical guidelines.

INTERVENTIONS:
Drug: Intravenous tirofiban combination therapy — Patients will enter the tirofiban treatment protocol immediately within half an hour after randomization and prior to the femoral artery puncture. Tirofiban is administered as an intravenous bolus dose of 10 μg/kg injection within 3 min and then by an intravenous infusion at a rate of 0.1 μg/(kg·min) for 24 hours.
  Other Names: Tirofiban
  Arms: Intervention group

SUMMARY:
In recent years, the positive results of trials for mechanical thrombectomy (MT) have brought a new era for large artery occlusion patients, especially those beyond the time window of intravenous thrombolysis. However, interventional procedures can cause endothelial injuries leading to local activation of platelet aggregation and subsequent thromboembolic complications or early re-occlusion.Tirofiban is a specific antagonist of the platelet glycoprotein (GP) IIb/IIIa receptor, which is considered highly effective against the final common pathway of platelet aggregation and preventing vascular reocclusion. However, there is no consensus on if AIS patients treated with MT also benefit from intravenous tirofiban. This study aims to evaluate the effectiveness and safety of profiles of tirofiban during MT and provide reliable clinical evidence for the treatment of tirofiban in AIS patients.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, open-label, randomized controlled, blinded-endpoint trial with two parallel groups and a 3-month follow-up. A total of 200 eligible participants recruited from 4-6 stroke centers will be randomly allocated to either an experimental group (intravenous tirofiban + MT therapy) or a control group (MT alone) in a 1:1 ratio. The primary outcome is a composite endpoint, including the rate of recanalisation after the first embolectomy and the risk of symptomatic intracerebral haemorrhage. The secondary outcomes include clinical and neuroimaging outcomes, procedure-related complications, and adverse events to evaluate the effects of MT in combination with tirofiban treatment compared to MT alone in AIS patients. Intention-to-treat (ITT) analysis will be undertaken in this study, and the full analysis set (FAS) population serves as the primary population for the analysis of efficacy data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years (including 18 and 85);
2. Acute ischemic stroke within 24 hours of onset, and NIHSS >5 points;
3. Acute large vessel occlusion, including internal carotid artery, M1 segment of middle cerebral artery, M2 segment of middle cerebral artery;
4. Multimodal CT/MRI imaging was completed before thrombectomy, and the following criteria were met: penumbra>10ml, infarct core volume <70ml, and mismatch rate >1.2;
5. Planned to receive endovascular treatment;
6. Informed consent was obtained.

Exclusion Criteria:

1. History of atrial fibrillation or atrial flutter, or 12-lead ECG before randomization and after admission showing atrial flutter or atrial fibrillation;
2. Treated with intravenous thrombolysis for this stroke or currently taking new oral anticoagulant drugs, warfarin, ticagrelor and other drugs that may increase the risk of bleeding;
3. Pre-stroke disability (pre-stroke mRS score > 2);
4. Severe comorbidity (such as severe cardiopulmonary dysfunction, or the terminal stage of malignant tumors with expected survival less than 90 days);
5. CT shows hypodensity lesions in more than 1/3 of the territory of the middle cerebral artery;
6. Allergy to tirofiban or having any contraindications to the use of tirofiban (patients with active internal bleeding, history of intracranial hemorrhage, intracranial tumors, arteriovenous malformations, and intracranial aneurysms, or patients resulting in thrombocytopenia from the use of tirofiban previously);
7. Contraindications to the contrast agents used in multimodal CT/MRI examination (such as allergy to the contrast agents, etc.);
8. Pregnant or breastfeeding women;
9. Patients currently participating in other clinical study trials;
10. Other conditions determined by the investigator are not suitable for inclusion in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2023-07-08 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Composite rates of target vessel revascularization and no symptomatic intracerebral haemorrhage | 24-72hours after thrombectomy;
  Target vessel revascularization is defined as a modified thrombolysis in cerebral infarction (mTICI) grade after onepass thrombectomy procedure over grade 2b. Symptomatic intracerebral haemorrhage is defined according to per Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST) criteria.

SECONDARY OUTCOMES:
Recanalisation rates of the target vessel | 24-72 hours after thrombectomy;
  Neuroimaging outcomes
Dichotomized mRS score/ ordinal mRS score | The 90-day after randomisation
  Functional prognosis of the patient，clinical outcomes
Symptomatic intracerebral haemorrhage | By the end of the 90-day follow-up
  procedure-related complications and adverse events
Death | By the end of the 90-day follow-up
  procedure-related complications and adverse events
The number of thrombectomy times | By the end of the 90-day follow-up
  Treatment information

CONTACTS AND LOCATIONS:
Overall Officials: Gang Li, Principal Investigator — Shanghai East Hospital
Locations (1):
- Gang Li, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Background] Nogueira RG, Jadhav AP, Haussen DC, Bonafe A, Budzik RF, Bhuva P, Yavagal DR, Ribo M, Cognard C, Hanel RA, Sila CA, Hassan AE, Millan M, Levy EI, Mitchell P, Chen M, English JD, Shah QA, Silver FL, Pereira VM, Mehta BP, Baxter BW, Abraham MG, Cardona P, Veznedaroglu E, Hellinger FR, Feng L, Kirmani JF, Lopes DK, Jankowitz BT, Frankel MR, Costalat V, Vora NA, Yoo AJ, Malik AM, Furlan AJ, Rubiera M, Aghaebrahim A, Olivot JM, Tekle WG, Shields R, Graves T, Lewis RJ, Smith WS, Liebeskind DS, Saver JL, Jovin TG; DAWN Trial Investigators. Thrombectomy 6 to 24 Hours after Stroke with a Mismatch between Deficit and Infarct. N Engl J Med. 2018 Jan 4;378(1):11-21. doi: 10.1056/NEJMoa1706442. Epub 2017 Nov 11. PMID 29129157
- [Background] Albers GW, Marks MP, Kemp S, Christensen S, Tsai JP, Ortega-Gutierrez S, McTaggart RA, Torbey MT, Kim-Tenser M, Leslie-Mazwi T, Sarraj A, Kasner SE, Ansari SA, Yeatts SD, Hamilton S, Mlynash M, Heit JJ, Zaharchuk G, Kim S, Carrozzella J, Palesch YY, Demchuk AM, Bammer R, Lavori PW, Broderick JP, Lansberg MG; DEFUSE 3 Investigators. Thrombectomy for Stroke at 6 to 16 Hours with Selection by Perfusion Imaging. N Engl J Med. 2018 Feb 22;378(8):708-718. doi: 10.1056/NEJMoa1713973. Epub 2018 Jan 24. PMID 29364767
- [Background] Kellert L, Hametner C, Rohde S, Bendszus M, Hacke W, Ringleb P, Stampfl S. Endovascular stroke therapy: tirofiban is associated with risk of fatal intracerebral hemorrhage and poor outcome. Stroke. 2013 May;44(5):1453-5. doi: 10.1161/STROKEAHA.111.000502. Epub 2013 Mar 5. PMID 23463755
- [Background] Teng D, Pannell JS, Rennert RC, Li J, Li YS, Wong VW, Chien S, Khalessi AA. Endothelial trauma from mechanical thrombectomy in acute stroke: in vitro live-cell platform with animal validation. Stroke. 2015 Apr;46(4):1099-106. doi: 10.1161/STROKEAHA.114.007494. Epub 2015 Feb 24. PMID 25712942
- [Background] Muniz-Lozano A, Rollini F, Franchi F, Angiolillo DJ. Update on platelet glycoprotein IIb/IIIa inhibitors: recommendations for clinical practice. Ther Adv Cardiovasc Dis. 2013 Aug;7(4):197-213. doi: 10.1177/1753944713487781. Epub 2013 Jul 1. PMID 23818658
- [Background] Yang J, Wu Y, Gao X, Bivard A, Levi CR, Parsons MW, Lin L; INSPIRE Study Groupdagger. Intraarterial Versus Intravenous Tirofiban as an Adjunct to Endovascular Thrombectomy for Acute Ischemic Stroke. Stroke. 2020 Oct;51(10):2925-2933. doi: 10.1161/STROKEAHA.120.029994. Epub 2020 Sep 16. PMID 32933416
- [Background] Yang M, Huo X, Gao F, Wang A, Ma N, Shi H, Chen W, Wang S, Wang Y, Miao Z. Low-dose rescue tirofiban in mechanical thrombectomy for acute cerebral large-artery occlusion. Eur J Neurol. 2020 Jun;27(6):1056-1061. doi: 10.1111/ene.14170. Epub 2020 Mar 17. PMID 32048389
- [Background] Neuberger U, Seker F, Schonenberger S, Nagel S, Ringleb PA, Bendszus M, Pfaff JAR, Mohlenbruch MA. Prediction of intracranial hemorrhages after mechanical thrombectomy of basilar artery occlusion. J Neurointerv Surg. 2019 Dec;11(12):1181-1186. doi: 10.1136/neurintsurg-2019-014939. Epub 2019 Jun 1. PMID 31154353
- [Background] Wu Y, Yin C, Yang J, Jiang L, Parsons MW, Lin L. Endovascular Thrombectomy. Stroke. 2018 Nov;49(11):2783-2785. doi: 10.1161/STROKEAHA.118.022919. PMID 30355186
- [Background] Guo Y, Lin Y, Tang Y, Tang Q, Wang X, Pan X, Zou J, Yang J. Safety and efficacy of early antiplatelet therapy in acute ischemic stroke patients receiving endovascular treatment: A systematic review and meta-analysis. J Clin Neurosci. 2019 Aug;66:45-50. doi: 10.1016/j.jocn.2019.05.028. Epub 2019 May 29. PMID 31153752
- [Background] Zhou J, Gao Y, Ma QL. Safety and efficacy of tirofiban in acute ischemic stroke patients not receiving endovascular treatment: a systematic review and meta-analysis. Eur Rev Med Pharmacol Sci. 2020 Feb;24(3):1492-1503. doi: 10.26355/eurrev_202002_20208. PMID 32096199
- [Background] Sun Y, Guo ZN, Yan X, Wang M, Zhang P, Qin H, Wang Y, Zhu H, Yang Y. Safety and efficacy of tirofiban combined with endovascular therapy compared with endovascular therapy alone in acute ischemic stroke: a meta-analysis. Neuroradiology. 2021 Jan;63(1):17-25. doi: 10.1007/s00234-020-02530-9. Epub 2020 Aug 25. PMID 32844236
- [Derived] Lin L, Liu F, Yi T, Zhu Y, Yang J, Zhao Y, Wang F, Xiang G, Chen C, Xiao Y, Shen H, Xu L, Long Y, Zhang Y, Huang Z, Chen C, Churilov L, Parsons MW, Chen W, Li G; OPTIMISTIC Investigators. Tirofiban on First-Pass Recanalization in Acute Stroke Endovascular Thrombectomy: The OPTIMISTIC Randomized Clinical Trial. JAMA Netw Open. 2025 Apr 1;8(4):e255308. doi: 10.1001/jamanetworkopen.2025.5308. PMID 40244586